CLINICAL TRIAL: NCT00343031
Title: Effect of the Antiandrogen DDE on Anthropometric Measures at Birth - Anogenital Distance
Brief Title: Effect of the Antiandrogen DDE on Anthropometric Measures at Birth
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901177; 01-E-N177
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12-10

CONDITIONS: DDT
Keywords: Insecticides; Children; Women; Infection; DDT; Contaminant
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant women delivering male infants: Male newborns and their mothers living in Tapachula (Chiapas, Mexico) and surrounding areas exposed to DDT through house spraying programs to control malaria, grouped by level of DDT exposure.

SUMMARY:
Experimental studies have documented the p'p-DDT, p'p-DDE (a metabolite of DDT) and other organochlorine (OC) compounds have estrogenic and/or antiandrogenic activities capable of altering normal endocrine functions. It has been postulated that exposure to these toxins during embriogenesis may cause urogenital malformations. However, this hypothesis has not yet been evaluated in humans populations with relatively high levels of exposure. The primary goal of this project is to study in utero exposure to DDE in relation to anogenital distance in humans. Anogenital distance is measured from a gender and species specific landmark on the genitalia, such as the junction of the penis and the scrotum in male humans, to the center of the anus. Altered anogenital distance is a sensitive manifestation of prenatal endocrine disruption in animal models; whether it is a sensitive endpoint in humans has not been studied. We will test the hypothesis that DDE, an androgen-receptor blocker, decreases anogenital distance in male humans who have been chronically but not occupationally exposed to DDT in Mexico. Study participants will be newborns and their mothers who live in the state of Chiapas, Mexico and who have been exposed to DDT through house spraying programs to control malaria in this area. Anogenital distance will be measured at birth and in utero exposure to DDE will be determined by measuring DDE in maternal blood.

Demonstration that p'p-DDT or p'p-DDE may interfere with normal endocrine functions during embriogenesis will provide a model to increase our understanding of how other- more prevalent-environmental estrogens may act and will open new possibilities for research and potential control of etiologic factors related with this important public health problem....

DETAILED DESCRIPTION:
We propose to follow the women and children enrolled in our original study (n= approximately 850 of each). In the original study, women were enrolled and interviewed while in the hospital for delivery, their blood was drawn, and anthropometric measurements were performed on their newborn male infants.

The follow-up will be done primarily to determine the number of months that the mother breast feeds her child. Secondary endpoints will be infant infection as reported by the mother, and child growth as determined by measurement of height and weight and related measures (none in the genital region, as in the original study). Breast feeding duration, infections, and growth may be related to exposure to the DDT metabolite, DDE.

The follow-up visits will be every three months from 6 to 18 months after birth, and study nurses will visit subjects in their home. For some subjects, there would be fewer follow-up visits, due to study scheduling or breastfeeding cessation.

Mothers would be interviewed and mothers and children will undergo standard anthropometric assessments. This protocol does not call for collection of biologic specimens and poses minimal risk to subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pregnant women delivering male infants in Tapachula and surrounding areas.

EXCLUSION CRITERIA:

Women must not be over 35 years of age.

A physician's diagnosis of multiple fetuses, pre-eclampsia or pregnancy-related hypertension disorders or psychiatric, kidney, or cardiac disease; gestational diabetes; history of repeated urinary infections; seizure disorder requiring daily medications; ingestion of corticosteroids, and non-Spanish speakers.

At time of birth, additional exclusion criteria will include: an Apgar score (at five minutes) of 6 or less; any condition requiring treatment in the neonatal intensive care unit.

Infants must not have any condition requiring treatment in the neonatal intensive care unit.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2118 (Actual)
Dates: Start 2001-05-14; Study Completion 2019-12-10

PRIMARY OUTCOMES:
Child growth as determined by measurement of height and weight and related measures | Every 3 months from 6 to 18 months after birth
  Anogenital distance in male infants

SECONDARY OUTCOMES:
Number of months the mother breast fed her child | every 3 months from 6 to 18 months after birth
  Duration of breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Taneja, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institute for Public Health, Cuernavaca, Mexico

REFERENCES:
- [Background] Gilmore HT, Milroy M, Mello BJ. Supernumerary nipples and accessory breast tissue. S D J Med. 1996 May;49(5):149-51. PMID 8936016
- [Background] Callegari C, Everett S, Ross M, Brasel JA. Anogenital ratio: measure of fetal virilization in premature and full-term newborn infants. J Pediatr. 1987 Aug;111(2):240-3. doi: 10.1016/s0022-3476(87)80075-6. PMID 3612396
- [Background] Boklage CE. Interactions between opposite-sex dizygotic fetuses and the assumptions of Weinberg difference method epidemiology. Am J Hum Genet. 1985 May;37(3):591-605. PMID 4039888